CLINICAL TRIAL: NCT03414528
Title: Towards Identification of New Inborn Errors of Immunity by Whole Exome/Genome Sequencing
Brief Title: Identification of New Inborn Errors of Immunity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Janine Reichenbach, Co-Head Division Immunology, University of Zurich
Other Study IDs: Ident_PID
Record Dates: First submitted 2018-01-10; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Primary Immune Deficiency Disorder
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with PID
  Interventions: Diagnostic Test: Diagnostic Test

INTERVENTIONS:
Diagnostic Test: Diagnostic Test — Analysis of DNA samples of patients with molecularly undetermined PID by whole exome/genome sequencing Transcriptome analysis of patients with molecularly undetermined PID

SUMMARY:
Analysis of DNA samples of patients with molecularly undetermined PID by whole exome/genome sequencing.

Transcriptome analysis of patients with molecularly undetermined PID.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary immunodeficiency (PID)
* Male and Female participants 0 years to adult age (any)
* Written informed consent by the participant after information about the research project

Exclusion Criteria:

* Secondary immunodeficiency
* Refusal to enter the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with unidentified inborn error of immunity (primary immunodeficiency, PID) or optionally healthy direct relatives, to determine whether they are carriers of the disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-08-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Identification of the genetic defects | 10 years
  Whole exome/Genome sequencing will be done to identify new mutations leading to immunodeficiency

CONTACTS AND LOCATIONS:
Overall Officials: Janine Reichenbach, Prof. Dr., Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
We are planning to share IPD in the form of Scientific publications in peer-reveiwed journals and communications at Scientific meetings